CLINICAL TRIAL: NCT00294112
Title: A Phase II, Open-label, Randomized Study to Evaluate the Safety and Efficacy of PROCHYMAL™ IBD (ex Vivo Cultured Adult Human Mesenchymal Stem Cells) Intravenous Infusion for the Treatment of Subjects Experiencing Moderate-to-severe Crohn's Disease That is Refractory to Steroids and Immune Suppressants
Brief Title: Prochymal™ Adult Human Mesenchymal Stem Cells for Treatment of Moderate-to-severe Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mesoblast, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSIRIS-601-602
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Crohn's Disease
Keywords: mesenchymal stem cells
MeSH Terms: conditions — Crohn Disease | interventions — remestemcel-l

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High dose (Experimental): High dose (8 million cells per kg of body weight)
  Interventions: Drug: Prochymal™ adult human mesenchymal stem cells; Drug: adult human mesenchymal stem cells
- Low dose (Experimental): Low dose: 2 million cells per kg body weight
  Interventions: Drug: Prochymal™ adult human mesenchymal stem cells; Drug: adult human mesenchymal stem cells

INTERVENTIONS:
Drug: Prochymal™ adult human mesenchymal stem cells — Cells in plasmalyte and containing dimethylsulfoxide
  Other Names: PROCHYMAL
Drug: adult human mesenchymal stem cells — two infusions, one week apart, each comprising adult human mesenchymal stem cells
  Other Names: PROCHYMAL

SUMMARY:
Human mesenchymal stem cells (MSCs), derived from healthy adult volunteer human donors, can be obtained from bone marrow donation and cultured in the laboratory. MSCs have shown the ability to find injured tissue, reduce and control inflammation, and assist in tissue repair.

Prochymal™ MSCs will be infused into patients with moderate-to-severe Crohn's disease. Infusions will occur on two separate days, 7-10 days apart. Patients will be monitored for reduced Crohn's disease symptoms.

DETAILED DESCRIPTION:
Human mesenchymal stem cells (MSCs), derived from healthy adult volunteer human donors, can be obtained from bone marrow donation and cultured in the laboratory. MSCs have shown the ability to find injured tissue, reduce and control inflammation, and assist in tissue repair.

Prochymal™ MSCs will be infused into patients with moderate-to-severe Crohn's disease. Infusions will occur on two separate days, 7-10 days apart. Patients will be monitored for reduced Crohn's disease symptoms. Patients will receive high or low dose. Study is open label.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18 to 70 years of age, inclusive.
2. If female and of child-bearing age, subject must be non-pregnant, non-breast-feeding, and use adequate contraception. If male, subject must use adequate contraception.
3. Subject must have endoscopically or radiographically active Crohn's disease
4. Subject must have a Crohn's disease activity index (CDAI) of at least 220.
5. Subject must have a C-reactive protein (CRP) of at least 5 mg/l.
6. Subject must have ileocolitis, colitis, or ileitis.
7. At some time during the course of the subject's Crohn's disease (CD), subject must have received both steroids and immunosuppressive agents (for example, azothioprine, 6-mercaptopurine, or methotrexate) which did not control the CD.
8. Subject may be receiving antibiotics, 5-aminosalicylic acid, azathioprine, 6-mercaptopurine, methotrexate, prednisone, or any similar drugs at the time of enrollment.

   * The dose of 5-aminosalicylic acid (5-ASA) must have been stable for at least 4 weeks prior to enrollment.
   * The dose of steroids must have been stable for at least 4 weeks prior to enrollment.
   * The dose of antibiotics must have been stable for at least 4 weeks prior to enrollment.
   * The dose of immunosuppressants (for example, azathioprine, 6-mercaptopurine [6-MP], or methotrexate) must have been stable for at least 8 weeks prior to enrollment and the subject on therapy for at least three months prior to enrollment.
9. Subject must have adequate renal function as defined by a calculated creatinine clearance of greater than 30 ml/min using the Cockcroft-Gault equation, and a serum creatinine concentration of less than 2.0 mg/dl.
10. Subject must be available for all specified assessments at the study site through day 30.
11. Subject must provide a written informed consent form (ICF) and authorization for use of and disclosure of personal health information (PHI).

Exclusion Criteria:

1. Subject has any alcohol or substance abuse within 6 months of randomization.
2. Subject has evidence of fibrostenotic obstructive Crohn's disease.
3. Subject has an active infection with HIV or hepatitis B or C.
4. Subject has had surgery or trauma within 28 d prior to enrollment.
5. Subject has a known allergy to computed tomography (CT) contrast agents.
6. Subject has a known allergy to bovine or porcine products.
7. Subject has body mass greater than 150 kg.
8. Subject has had a stricture of the bowel requiring hospitalization within 6 months prior to enrollment.
9. Subject has had bowel surgery other than perianal (for example, fistulotomy, seton placement, or abscess drainage) within 6 months prior to enrollment.
10. Subject has received infliximab; adalimumab; or other antibody, protein, or biological therapy not specifically approved by the United States Food and Drug Administration (FDA) for Crohn's disease for 90 days (d) prior to enrollment in study.
11. Subject has received prednisone greater than 20 mg/d at any time 28 d prior to enrollment in study.
12. Subject has a permanent colostomy or ileostomy.
13. Subject has aspartate aminotransferase (AST), alkaline phosphatase (ALP), or alanine transaminase (ALT) more than 2.5 times the upper limit of normal at screening.
14. Subject has evidence of active malignancy other than resected basal or squamous cell carcinoma of the skin, or prior history of active malignancy that has not been in remission for at least 5 years.
15. Subject has history of bacteremia or other serious bacterial or fungal infection in past 3 months other than a treated urinary tract infection or drained perianal abscess.
16. Subject has received an investigational agent (IA)-an agent or device not approved by FDA for marketed use in any indication-within 90 d (or 5 half-lives, whichever is longer) of randomization.
17. Subject has cardiopulmonary disease that, in the opinion of the Investigator, is either unstable or severe enough to justify exclusion from this study.
18. Subject has any underlying or current medical or psychiatric condition that, in the opinion of the Investigator, would make participation in the study unsafe.
19. Subject has any underlying or current medical or psychiatric condition that, in the opinion of the Investigator, would interfere with the evaluation of the subject. Such excluding conditions might include, for example, uncontrolled infection, right heart failure, pulmonary hypertension.
20. Subject has unstable arrhythmia.
21. Subject is unwilling or unable to adhere to requirements of protocols.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-03-13 (Actual); Primary Completion 2006-07-21 (Actual); Study Completion 2006-07-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Reduction in Crohn's Disease Activity Index (CDAI) of at Least 100 Points | 28 days
  The CDAI is a composite index of 8 disease variables (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations or fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight). Scores range from approximately 0 to 600, with a higher score indicating more disease activity.

SECONDARY OUTCOMES:
Number of Participants with Reduction in CDAI of at Least 70 points | 28 days
  The CDAI is a composite index of 8 disease variables (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations or fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight). Scores range from approximately 0 to 600, with a higher score indicating more disease activity.
Improvement as Assessed by the Inflammatory Bowel Disease Questionnaire (IBDQ) | 28 days
  The IBDQ measures disease-specific quality of life by assessing bowel symptoms, systemic symptoms, emotional function, and social function. Subscores can range from 1 (worst) to 7 (best). The total IBDQ is calculated as the sum of the responses to the individual IBDQ questions. The total score ranges from 32 to 224. An increase in score from baseline indicates improvement.
Time to Improvement in IBDQ | 28 days
Number of Participants with Reduction of at Least 50% in Fistulas in Participants with Fistulas Draining Under Moderate Compression | 28 days
Number of Participants with Induction of Remission as Defined by Reduction of CDAI to Below 150 | 28 days
  The CDAI is a composite index of 8 disease variables (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations or fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight). Scores range from approximately 0 to 600, with a higher score indicating more disease activity.
Time to Reduction in CDAI of at Least 100 Points | 28 days
Time to Reduction in CDAI of at Least 70 Points | 28 days
Time to Induction of Remission as Defined by Reduction of CDAI to Below 150. | 28 days
Number of Participants with Adverse Events | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mahboob Rahman, MD, Study Director — Mesoblast, Inc.
Locations (4):
- United States (4):
  - Osiris Clinical Site, Baton Rouge, Louisiana
  - Osiris Clinical Site, Charlotte, North Carolina
  - Osiris Clinical Site, Pittsburgh, Pennsylvania
  - Osiris Clinical Site, Richmond, Virginia